CLINICAL TRIAL: NCT06086379
Title: Cognitive Rehabilitation to Improve Functioning in Veterans Following COVID-19
Brief Title: Cognitive Rehabilitation Therapy for COVID-19
Acronym: CCT-COVID
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E4764-W
Record Dates: First submitted 2023-10-13; First posted 2023-10-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: Post-Acute COVID-19 Syndrome; Cognitive rehabilitation; Cognitive training; Cognitive remediation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — HCE

STUDY DESIGN:
Intervention Model Description: Two group randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CCT-C (Experimental): 10-week Compensatory Cognitive Training Group
  Interventions: Behavioral: Compensatory Cognitive Training for COVID-19
- HCE (Active Comparator): 10-week Holistic Cognitive Education Group
  Interventions: Behavioral: Holistic Cognitive Education

INTERVENTIONS:
Behavioral: Compensatory Cognitive Training for COVID-19 — CCT-C is a manualized group-based behavioral intervention (10 weeks, 2 hours per week, 20 hours total) designed to improve cognition and everyday functioning in patients with prolonged COVID-19 symptoms
  Other Names: CCT-C
  Arms: CCT-C
Behavioral: Holistic Cognitive Education — HCE provides the same frequency and amount of therapist and other group member contact as CCT-C, but does not provide training in cognitive or lifestyle strategies addressed in CCT-C. The HCE intervention provides information and discussion regarding common causes of and treatments for cognitive impairment.
  Other Names: HCE
  Arms: HCE

SUMMARY:
Cognitive dysfunction, psychiatric symptoms, functional impairment, and disability following COVID-19 negatively impact Veterans' community functioning and quality of life, contribute to significant human suffering, and are costly to VHA. Rehabilitation is a critical priority for Veterans with long COVID. One promising treatment to improve functioning in Veterans with post-COVID-19 cognitive symptoms is Compensatory Cognitive Training (CCT). Previous studies have found that CCT is feasible, acceptable, and efficacious in Veteran populations with multiple sources of cognitive dysfunction. This randomized controlled trial aims to address important RR&D priorities by examining feasibility, acceptability, and preliminary efficacy of a COVID-19-specific rehabilitation intervention, CCT for long COVID (CCT-C) compared to a robust control condition. The proposed study has the potential to improve cognitive function, functional independence, and quality of life for Veterans with late or delayed effects of secondary conditions related to COVID-19 infections.

DETAILED DESCRIPTION:
2-8% of the US population report "long COVID" symptoms - including "brain fog," thinking difficulties, memory problems, and psychiatric symptoms such as sleep disturbance, anxiety, and depression. Rates of post-COVID-19 symptoms are nearly double in the Veteran population. These cognitive symptoms contribute to functional impairments, reduced quality of life, poorer self-reported health status, psychological distress, delayed return to work, new onset disability, reduced community integration, and increased healthcare utilization. One promising treatment to improve both everyday functioning and cognition secondary to post-COVID-19 symptoms is Compensatory Cognitive Training (CCT). Previous studies have found that CCT is feasible, acceptable, and efficacious in Veteran populations with multiple sources of cognitive dysfunction. The proposed CDA provides a golden opportunity to evaluate CCT for Veterans with prolonged COVID-19 symptoms (CCT-C), compared with a robust control condition, Holistic Cognitive Education (HCE). The project closely aligns with current RR&D priorities, by "examining COVID-19-specific rehabilitation interventions and responses to treatment" and by addressing "late or delayed effects of secondary conditions related to COVID-19 infections on impairment and disability." Specific aims are 1) to conduct a pilot randomized controlled trial of remote CCT-C with 70 Veterans (35 CCT-C, 35 HCE) with post-COVID-19 cognitive symptoms to examine feasibility, acceptability, and initial efficacy; 2) to examine the preliminary efficacy of CCT-C in this population on overall functioning, as measured by the World Health Organization's Disability Assessment Schedule (WHODAS 2.0), performance-based measures of functional capacity, and secondary outcomes (cognitive performance, quality of life, self-reported cognitive problems, psychiatric symptoms, sleep disturbance, and engagement in work/community activities); and 3) to explore moderators of outcome (e.g., age, initial COVID-19 severity, baseline cognitive functioning, presence of PTSD/mTBI history; biomarkers related to COVID-19 infection).

ELIGIBILITY:
Inclusion Criteria:

* Veterans > 18 years old who are able to provide informed consent
* Prior participation in SF Parent Study or LA Parent Study
* Report of cognitive symptoms that Veteran attributes to COVID-19 infection

Exclusion Criteria:

* Current substance abuse disorder, psychotic disorder, dementia, etc.
* History of moderate to severe brain injury with loss of consciousness > 30 minutes
* Auditory or visual impairments that would prevent the ability to participate in assessment procedures
* Invalid performance on one or more embedded performance validity tests (PVTs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in World Health Organization - Disability Assessment Schedule (WHODAS 2.0) | baseline, 8 weeks
  Change in average total score

SECONDARY OUTCOMES:
Change in objective cognitive performance z score | baseline, 8 weeks
  Change in composite z score
Change in functional capacity performance z score | baseline, 8 weeks
  Change in composite z score
Change in Patient Health Questionnaire 9 (PHQ-9) | baseline, 8 weeks
  Change in total score
Change in Generalized Anxiety Disorder 7 (GAD-7) | baseline, 8 weeks
  Change in total score
Change in PTSD Checklist for DSM-5 (PCL-5) | baseline, 8 weeks
  Change in total score
Change in Cognitive Failures Questionnaire (CFQ) | baseline, 8 weeks
  Change in total score
Change in Neuro-QOL: Applied Cognition General Concerns | baseline, 8 weeks
  Change in total score
Change in Neuro-QOL: Applied Cognition Executive Functioning | baseline, 8 weeks
  Change in total score
Change in Neuro-QOL: Fatigue | baseline, 8 weeks
  Change in total score
Change in World Health Organization - Quality of Life (WHOQOL-BREF) | baseline, 8 weeks
  Change in total score
Change in Insomnia Severity Index (ISI) | baseline, 8 weeks
  Change in total score

CONTACTS AND LOCATIONS:
Overall Officials: Tara A Austin, AA, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No